CLINICAL TRIAL: NCT02492386
Title: Safety and Feasibility of Bioabsorbable Everolimus-Eluting Stents for Patients With Internal Pudendal Artery-Related Arteriogenic Erectile Dysfunction (PERFECT-ABSORB)
Brief Title: Bioabsorbable Everolimus-Eluting Stents for Internal Pudendal Artery-Related Arteriogenic Erectile Dysfunction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201501059DIPB
Record Dates: First submitted 2015-06-24; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Impotence, Arteriogenic
Keywords: bioabsorbable vascular scaffold; erectile dysfunction
MeSH Terms: conditions — Impotence, Vasculogenic; Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Bioabsorbable everolimus-eluting stent deployment
  Interventions: Device: Bioabsorbable everolimus-eluting stent deployment

INTERVENTIONS:
Device: Bioabsorbable everolimus-eluting stent deployment — Bioabsorbable everolimus-eluting stent deployment

SUMMARY:
In this prospective, unblinded, single-arm, single-center study, investigators would like to assess the feasibility and safety of the bioabsorbable everolimus-eluting stents in patients with erectile dysfunction and concomitant internal pudendal artery stenoses. A total of 15 bioabsorbable vascular scaffolds (BVSs) are planned to be assessed and will be deployed in the internal pudendal artery, with a 1:1 ratio of both proximal and distal segments.

DETAILED DESCRIPTION:
Background: Obstructive pelvic arterial lesions were present in approximately 70-80% of patients aged >50 years and having erectile dysfunction. Previous studies have shown that most arterial stenoses were present in the internal pudendal and common penile artery segments. Investigators have also demonstrated that angioplasty for both internal pudendal and penile arteries is safe and can achieve clinically significant improvement in erectile function in ~60% of patients with erectile dysfunction. Nevertheless, in the ZEN study and investigators' preliminary observation, the 6-month angiographic binary restenosis rate for drug-eluting stents (DES) in internal pudendal artery approached 30-50%. The internal pudendal artery requires integral vasomotor function to provide sufficient blood supply during erection, whereas metallic stents impair vasomotor function. A fully bioabsorbable drug-eluting stent that scaffolds the vessel wall when needed and then disappear once the acute recoil and constrictive remodeling processes have subsided is therefore particularly advantageous for the internal pudendal artery. Investigators herein would like to assess the feasibility and safety of the bioabsorbable everolimus-eluting stents in patients with erectile dysfunction and concomitant internal pudendal artery stenoses.

Methods: This prospective, unblinded, single-arm, single-center study is a feasibility trial designed to provide preliminary observations and generate hypotheses for future studies. A total of 15 BVSs are planned to be assessed and will be deployed in the internal pudendal artery, with a 1:1 ratio of both proximal and distal segments. All subjects will undergo pelvic CT angiography at baseline and 6 months after intervention. Invasive selective pudendal angiography will be performed 6-9 months after intervention as well. Intravascular ultrasound and/or optical coherence tomography (OCT) imaging will be obtained during invasive angiography. The primary feasibility endpoint is CT angiographic binary restenosis (≥50% lumen diameter stenosis) at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* men 20 years of age or older with "consistent" erectile dysfunction defined as both IIEF-5 scores, taken at least 4 weeks apart, are in the range of 5 to 21 points and with a difference of ≤2 points;
* the anatomical inclusion criteria, based on pelvic CT angiography, are unilateral luminal diameter stenosis ≥70% or bilateral diameter stenoses ≥50% in the internal pudendal arteries with reference vessel diameter ≥2.5 mm and ≤4.0 mm and a target-lesion length ≤30 mm.

Exclusion Criteria:

* the arterial inflow to the penis is entirely from the accessory pudendal arteries rather than the usual internal pudendal artery and common penile artery;
* the presence of focal diameter stenosis ≥70% in the common penile artery, internal iliac artery, or anterior division of inferior gluteal artery;
* previous radical prostatectomy, pelvic radiation, or Peyronie's disease;
* untreated hypogonadism (serum total testosterone <300 ng/dL within 14 days before enrollment);
* acute coronary syndrome, stroke, or life-threatening arrhythmia within 3 months before enrollment;
* poorly controlled diabetes mellitus with glycosylated hemoglobin levels >9%;
* serum creatinine levels >2.5 mg/dL;
* bleeding diathesis or known hypercoagulopathy;
* life expectancy of fewer than 12 months;
* known intolerance to contrast agents.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-09 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
CT angiographic binary restenosis | 6 months
  Binary restenosis is defined as >=50% lumen diameter stenosis

SECONDARY OUTCOMES:
Diameter measured by invasive angiography | 6-9 months
  Diameter will be measured by invasive angiography at in-stent, peri-stent, and in-segment sections
Diameter stenosis measured by invasive angiography | 6-9 months
  Diameter stenosis will be measured by invasive angiography at in-stent, peri-stent, and in-segment sections
Late loss measured by invasive angiography | 6-9 months
  Late loss will be measured by invasive angiography at in-stent, peri-stent, and in-segment sections
International Index of Erectile Function (IIEF)-5 score | 1, 3, 6, and 12 months
Major adverse events | 1, 3, 6, and 12 months
  Major adverse events are defined as procedure-related death, occurrence of perineal hematoma, gangrene or necrosis (glans penis, penile shaft, scrotal, or anal), or the need for subsequent perineal, penile, or anal surgery (including target-lesion or vessel revascularization or arterial embolization procedures).

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Dau Wang, MD, PhD, Principal Investigator — Natioal Taiwan University Hospital

REFERENCES:
- [Background] Wang TD, Lee WJ, Yang SC, Lin PC, Tai HC, Hsieh JT, Liu SP, Huang CH, Chen WJ, Chen MF. Safety and six-month durability of angioplasty for isolated penile artery stenoses in patients with erectile dysfunction: a first-in-man study. EuroIntervention. 2014 May;10(1):147-56. doi: 10.4244/EIJV10I1A23. PMID 24832642